CLINICAL TRIAL: NCT00004250
Title: A Phase II Trial of Isolated Limb Infusion With Melphalan and Dactinomycin for Regional Melanoma and Soft Tissue Sarcoma of the Extremity
Brief Title: Isolated Limb Infusion of Chemotherapy in Treating Patients With Melanoma or Soft Tissue Sarcoma of the Arm or Leg That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 99-047; MSKCC-99047; NCI-G99-1664
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Melanoma (Skin); Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III melanoma; stage IV melanoma; recurrent melanoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Melanoma; Sarcoma | interventions — Dactinomycin; Melphalan

INTERVENTIONS:
Biological: dactinomycin
Drug: isolated limb perfusion
Drug: melphalan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Infusing chemotherapy to the tumor area only may kill more tumor cells and cause less damage to healthy tissues.

PURPOSE: This phase II trial is studying isolated limb infusion of chemotherapy to see how well it works in treating patients with melanoma or soft tissue sarcoma of the arm or leg that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of isolated limb infusion (ILI) with melphalan and dactinomycin in patients with primary or recurrent, unresectable regional melanoma or soft tissue sarcoma of the extremity.
* Determine the morbidity of patients treated with this regimen.
* Determine the expression of melanoma-associated antigens as well as cellular and humoral immune responses to these antigens in patients with regional disease.

OUTLINE: Patients undergo fluoroscopic placement of angiographic arterial and venous catheters into the appropriate extremity. After the limb is warmed, melphalan and dactinomycin are rapidly infused into the isolated limb via the arterial catheter. Melphalan and dactinomycin are then recirculated for 20 minutes. Patients with little or no response at 8 weeks may receive up to 2 additional treatments at the discretion of the treating physician.

Patients are followed at 1-2 weeks, 3-4 weeks, 6-8 weeks, and then every 3-6 months thereafter as deemed necessary by the treating physician.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primary or recurrent, regional melanoma or soft tissue sarcoma that is not amenable to surgical resection

  * Majority (greater than 95%) of disease must be distal to the apex of the femoral triangle in the lower limb and the deltoid insertion in the upper limb
* Bidimensionally measurable disease in the extremity
* Patients with disease beyond the limb are eligible if their extremity disease requires palliative treatment in the judgment of their physician

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 3,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* Must have palpable femoral/axillary, dorsalis pedis/popliteal, or radial pulses in the extremity to be treated
* No signs or symptoms of vascular insufficiency (no history of claudication or other ischemic peripheral vascular disease)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No other concurrent serious illness
* No severe diabetes

  * No prior extremity complications due to diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior antitumor therapy and recovered
* At least 2 weeks since prior antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 1999-08; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy
Morbidity
Expression of melanoma-associated antigens

CONTACTS AND LOCATIONS:
Overall Officials: Mary S. Brady, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Brady MS, Brown K, Patel A, Fisher C, Marx W. Isolated limb infusion with melphalan and dactinomycin for regional melanoma and soft-tissue sarcoma of the extremity: final report of a phase II clinical trial. Melanoma Res. 2009 Apr;19(2):106-11. doi: 10.1097/CMR.0b013e32832985e3. PMID 19282789